CLINICAL TRIAL: NCT06626152
Title: Measuring Psychomotor Response to L-DOPA Challenge As a Biomarker for Outcomes in Late-Life Depression: a Pilot Feasibility Trial
Acronym: LLDOPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Providence Health & Services (Other)
Responsible Party: Principal Investigator, Kevin Smith, Clinical Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLDOPA
Record Dates: First submitted 2024-09-03; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- L-DOPA Challenge (Experimental): Participants will be administered a levodopa-carbidopa challenge, at a dosage of 150mg/37.5mg once daily for one week, followed by twice daily for one week. Psychomotor speed will be assessed before and after the challenge.
  Interventions: Drug: Apo-levocarb

INTERVENTIONS:
Drug: Apo-levocarb — As above.

SUMMARY:
Background

Adults over the age of 60 with symptoms of major depressive disorder are said to have late-life depression (LLD), a condition that usually decreases a person's quality of life and is associated with other risks like physical frailty and dementia. A common feature of more severe LLD is psychomotor slowing, where a person's ability to think and move are impaired. For example, they might not be able to walk or process information as quickly, and they might have problems with their working memory.

Psychomotor slowing in LLD might be the result of a problem with the way a person's body produces or responds to the neurotransmitter dopamine. The drug Levodopa (L-DOPA), which can replace missing dopamine in the brain, has been used to treat to treat Parkinson's disease for many decades, and it might also affect psychomotor slowing in LLD.

Methods

In this study, participants are adults aged 60 years or older with moderate to severe major depression. Participants undergo the "L-DOPA challenge"-a 2-week period where they receive a dose of L-DOPA once a day for the first week and a dose of L-DOPA twice a day for the second week. Before and after a participant completes the L-DOPA challenge, the study team assesses their depressive symptoms and psychomotor function. After the L-DOPA challenge, if a participant still shows signs of moderate or severe depression, they receive an antidepressant for 12 weeks.

Aims

The first aim of this study is to test the feasibility of the L-DOPA challenge-that is, whether most of the 50 participants recruited for this study will complete the L-DOPA challenge. For example, participants might have to withdraw if they can't make the daily visits to the research site to receive their L-DOPA medication, if they can't tolerate the medication's side effects, or if their depressive symptoms get significantly worse. Our hypothesis is that 80% of the participants will complete the L-DOPA challenge.

The second aim of the study is to see if L-DOPA affects participants' depressive symptoms, processing speed, and working memory. Our hypothesis is that L-DOPA response, measured as an improvement in gait speed, is associated with a decrease in depressive symptoms and an increase in processing speed and working memory.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient persons capable of providing informed consent
* Minimum age of 60 years old
* MINI International Neuropsychiatric Interview diagnosis of major depressive disorder, based on DSM-5 criteria
* MADRS score of ≥15 (moderate/severe depression)
* On stable doses of psychotropic medication, including antidepressant medication, for at least 4 weeks
* Able to adhere to the intervention schedule

Exclusion Criteria:

* Current diagnosis of major neurocognitive disorder
* Current active psychosis
* Unstable medical illness, including clinical or laboratory evidence of uncompensated cardiovascular, endocrine, hematologic, hepatic, pulmonary (including bronchial asthma), or renal disease
* Diagnosis of narrow angle glaucoma
* Suspicious, undiagnosed skin lesions or a history of melanoma
* History of myocardial infarction
* Atrial, nodal, or ventricular arrhythmias
* History of seizures or seizure disorder
* History of peptic ulcer disease
* History of allergy or other hypersensitivity to levodopa, carbidopa, or to any other ingredient in the formulation of Levocarb
* Active suicidal ideation
* Psychotropic medication initiation or dose change <4 weeks prior to enrolment
* Regular use of dopamine antagonist or benzodiazepines ≥2mg lorazepam equivalent per day
* Unable to complete neuropsychological testing in the English language
* Have a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests)
* History of falls, with ≥1 fall per week during the past 4 weeks

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
L-DOPA challenge completion rate | 6 months
  Number of participants who complete the 2-week challenge of receiving L-DOPA and post-challenge assessments
Depressive symptoms | At 2, 3, 7, and 15 weeks from baseline
  Change in depressive symptoms, as measured by the Montgomery-Åsberg Depression Rating Scale, after the L-DOPA challenge and after treatment for depression
Gait speed | At baseline and 2 weeks from baseline
  Change in gait speed in response to L-DOPA, as measured by time to complete the 4-metre walk test.
Psychomotor speed | At baseline and 2 weeks from baseline
  Changes in psychomotor speed in response to L-DOPA, as measured by the clinician-rated CORE instrument

SECONDARY OUTCOMES:
Processing speed | At 2 and 15 weeks from baseline
  Change in processing speed, as measured by the NIH Toolbox Cognitive Battery: Pattern Comparison tool, after the L-DOPA challenge and after treatment for depression
Working memory | At 2 and 15 weeks from baseline
  Change in working memory, as measured by the NIH Toolbox Cognitive Battery: List Sorting tool, after the L-DOPA challenge and after treatment for depression
Side effects related to L-DOPA | At 2 weeks from baseline
  Incidence, frequency, and severity of side effects following L-DOPA administration, related to the cardiovascular, respiratory, musculoskeletal, genitourinary, skin, and central nervous systems, as recorded on an Adverse Effects Monitoring Form

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada